CLINICAL TRIAL: NCT05415644
Title: Study of the Bioequivalence and Food Effects of HRX0701 Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRX0701-101
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: HRX0701 tablets are used alone, or Retagliptin phosphate tablets are used in combination with metformin hydrochloride tablets.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioequivalence study part (Experimental)
  Interventions: Drug: hrx0701 tablets、Metformin hydrochloride tablets、Retagliptin phosphate tablets
- Food impact study part (Experimental)
  Interventions: Drug: hrx0701 tablets

INTERVENTIONS:
Drug: hrx0701 tablets、Metformin hydrochloride tablets、Retagliptin phosphate tablets — High-specification group: subject preparation: HRX0701 (50 mg/1000 mg) 1 tablet (to be taken after a meal); Reference preparation: 1 tablet of retagliptin phosphate (50 mg), 2 tablets of metformin hydrochloride (Glucophage®) (500 mg), taken twice after meals.
  Low Specification Group:
  Preparation: HRX0701 (50 mg/850 mg) 1 tablet (taken after a meal); Reference: 1 tablet of retagliptin phosphate (50 mg), 1 tablet of metformin hydrochloride (Glucophage®) (850 mg), taken twice after meals.
  Arms: Bioequivalence study part
Drug: hrx0701 tablets — High specification group HRX0701 (FDC) tablets (50 mg / 1000 mg) for a total of 2 tablets (take 1 tablet after meals or on an empty stomach).
  Low-spec group HRX0701 (FDC) tablets (50 mg / 850 mg) for a total of 2 tablets (take 1 tablet after meals or on an empty stomach).
  Arms: Food impact study part

SUMMARY:
To evaluate the bioequivalence of a single oral dose of HRX0701 tablets and the reference formulations retagliptin phosphate tablets and metformin hydrochloride tablets in healthy subjects in the postprandial state; To evaluate the pharmacokinetic effects of a high-fat diet on retagliptin and metformin after a single oral administration of HRX0701 tablets in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 to 45 years (both ends of the value, subject to the signing of informed consent).
2. Male weight ≥ 50.0 kg, female weight ≥ 45.0 kg, and body mass index (BMI): 19~26 kg/m2 (including both ends).
3. Based on medical history, comprehensive physical examination, laboratory tests, 12-lead ECG, chest x-ray, vital signs, etc., the researchers determined that the subjects met the health criteria.
4. Voluntarily sign an informed consent form prior to the commencement of activities related to this trial, be able to understand the procedures and methods of this trial, and be willing to complete this trial in strict compliance with the clinical trial protocol.

Exclusion Criteria:

1. Have a history of any clinically serious disease or a disease or condition that the researcher believes may affect the results of the test, including but not limited to circulatory system, endocrine system, nervous system, digestive system, urinary system or blood, immune, psychiatric and metabolic disease history.
2. People with allergies, including those who are explicitly allergic to the research drug or any ingredient in the research drug, allergic to any food ingredients or have special requirements for diet, and cannot comply with the unified diet.
3. Those who have undergone any surgery within 3 months before screening, or who have not recovered after surgery, or who may have surgery or hospitalization plans during the estimated trial period.
4. Have taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines or dietary supplements within 2 weeks before the screening period;
5. Those who have consumed grapefruit or fruit juice products within 2 days before administration, any food or beverage containing caffeine (such as coffee, tea, chocolate, cola or other carbonated drinks containing caffeine, etc.), xanthine foods or alcohol.
6. The researcher determines that the subject has a medical condition that affects the absorption, distribution, metabolism and excretion of the drug or can reduce compliance or the researcher deems inappropriate.
7. Screening those who have participated in clinical trials of any drug or medical device within 3 months before screening.
8. Those who donated blood (or lost blood) within 3 months before screening and donated blood (or lost blood) ≥ 400 mL, or received blood transfusions.
9. Those who plan to receive live (attenuated) vaccines during the trial.
10. Have a birth plan at the end of the screening to follow-up period, or refuse to use medically approved contraception.
11. Smokers (average of 5 cigarettes or more per day).
12. An average daily intake of more than 25 g of alcohol in the 1 month prior to screening (e.g., 750 mL of beer, 250 mL of wine, or 50 mL of low-grade liquor);
13. Drug abusers or drug urine screening test positive.
14. Positive for hepatitis B surface antigen (HBsAg) within 1 month before screening or screening period, or positive for anti-hepatitis C virus (HCV), or positive for human immunodeficiency virus (HIV), or positive for syphilis antibody.
15. 12-lead electrocardiogram (ECG) shows abnormalities and is of clinical significance.
16. There are any abnormal laboratory test values that are clinically significant by the researchers; (Note: For abnormal laboratory tests with clinical significance, if there is a clear and reasonable reason, the retest can be retested within one week, and the retest results can be used to determine whether the subject meets the conditions).
17. Subjects may not be able to complete this study for other reasons or those whom the researchers believe should not be included.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
PK parameters Cmax, in the postprandial plasma of subjects in postprandial plasma | day 1 to day 18
PK parameters AUC0-t in the postprandial plasma of subjects in postprandial plasma | day 1 to day 18
PK parameters AUC0-∞ in the postprandial plasma of subjects in postprandial plasma | day 1 to day 18
The PK parameters of retagliptin and metformin in the blood plasma on fasting and after meals reach peak time (Tmax) | day 1 to day 18
The PK parameters of retagliptin and metformin in the blood plasma on fasting and after meals peak concentration (Cmax) | day 1 to day 18
The PK parameters of retagliptin and metformin in the blood plasma on fasting and after meals area under the drug-time curve (AUC0-t) | day 1 to day 18
The PK parameters of retagliptin and metformin in the blood plasma on fasting and after meals area under the drug-time curve (AUC0-∞) | day 1 to day 18

SECONDARY OUTCOMES:
Apparent distribution volume (Vz/F) | day 1 to day 18
apparent clearance (CL/F) | day 1 to day 18
terminal phase half-life (t1/2) | day 1 to day 18
retagliptin and metformin in plasma on fasting and after meals | day 1 to day 18
The main metabolites of retagliptin acid PK parameters Cmax | day 1 to day 18
The main metabolites of retagliptin acid AUC0-t | day 1 to day 18
The main metabolites of retagliptin acid AUC0-∞ | day 1 to day 18
Adverse events | day 1 to day 25

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Third Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided